CLINICAL TRIAL: NCT04154605
Title: ClariFix Rhinitis Randomized Controlled Trial
Brief Title: ClariFix Rhinitis RCT
Acronym: CR RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Instruments (Industry)
Collaborators: North American Science Associates Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 4666-001
Record Dates: First submitted 2019-10-31; First posted 2019-11-06 (Actual); Results first posted 2021-09-20 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Chronic Rhinitis
Keywords: Cryotherapy; Cryoablation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to ClariFix or a sham procedure. After the 90-day visit, control participants may crossover to active ClariFix treatment, if they continue to meet enrollment criteria.
Who Masked: Participant
Masking Description: All participants will be blinded to treatment assignment from procedure through their 90-day visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ClariFix (Active Comparator): Cryotherapy of the nasal passages with the ClariFix device.
  Interventions: Device: ClariFix cryotherapy
- Sham (Sham Comparator): Sham cryotherapy of the nasal passages with the ClariFix device
  Interventions: Device: Sham ClariFix cryotherapy

INTERVENTIONS:
Device: ClariFix cryotherapy — Bilateral freeze ablation of nasal tissue using the ClariFix device.
  Arms: ClariFix
Device: Sham ClariFix cryotherapy — Bilateral sham ablation procedure using the ClariFix device.
  Other Names: Sham
  Arms: Sham

SUMMARY:
A randomized, sham-controlled, single-blind study of cryotherapy as a treatment for chronic rhinitis.

DETAILED DESCRIPTION:
A prospective, multicenter, randomized, sham-controlled, single-blind (participants) study to demonstrate the superiority of treatment with the ClariFix cryotherapy device for reducing symptoms when compared with a sham treatment in patients with chronic rhinitis. The ClariFix device is a Class II FDA-cleared medical device that is intended to be used as a cryosurgical tool for the destruction of unwanted tissue during surgical procedures, including in adults with chronic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥21 years of age.
2. Has been diagnosed with chronic nonallergic or allergic rhinitis.
3. Have moderate to severe symptoms of rhinorrhea (individual reflective Total Nasal Symptoms Score [rTNSS] symptom rating of 2 or 3), mild to severe symptoms of nasal congestion (individual rTNSS symptom rating of 1, 2, or 3), and a minimum total rTNSS of 4 (out of 12) at baseline.
4. Have an allergy test (by skin prick or intradermal testing or by validated in vitro tests for specific Immunoglobin E [IgE]) on file within 12 months of the baseline visit.
5. Be an appropriate candidate for bilateral ClariFix treatment performed under local anesthesia.
6. Be willing and able to comply with all study elements, as indicated by their written informed consent.
7. Be willing and able to comply with all study elements and provide written consent.

Exclusion Criteria:

1. Have clinically significant anatomic obstructions that in the investigator's opinion limit access to the posterior nose, including but not limited to severe septal deviation or perforation, nasal polyps, and/or sinonasal tumor.
2. Have had previous sinus or nasal surgery within 6 months of study enrollment.
3. Have previously undergone cryotherapy or other surgical interventions for rhinitis.
4. Have an active nasal or sinus infection.
5. Have rhinitis symptoms that are primarily due to seasonal allergies.
6. Have plans to (or otherwise anticipates the need to) undergo an ENT (ear, nose, throat) procedure concurrently or within 3 months after the study procedure.
7. Is on prescribed anticoagulants (eg, warfarin, Plavix) or 325 mg aspirin that cannot be discontinued before the procedure (81 mg aspirin and herbal supplements are acceptable).
8. Be unable to discontinue ipratropium bromide (IB) at least 14 days before baseline and through the 90-day follow-up visit.
9. Have a history of chronic epistaxis or experienced a significant epistaxis event (defined as epistaxis requiring medical intervention) in the past 3 months.
10. Have a history of rhinitis medicamentosa.
11. Have had previous head and/or neck irradiation.
12. Have an allergy or intolerance to local anesthetic agents.
13. Have cryoglobulinemia, paroxysmal cold hemoglobinuria, cold urticaria, Raynaud's disease, and/or open and/or infected wounds at or near the target tissue.
14. Have a neurological, medical, psychiatric condition, or social circumstance that would potentially increase risk, interfere with study participation, or confound interpretation of study data.
15. Be participating in another clinical research study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2025-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony DelSignore, MD, Principal Investigator — Ichan School of Medicine, Mount Sinai, New York, NY
Locations (1):
- ENT Associates of South Florida, Coral Springs, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ClariFix | Sham
Started | 68 | 65
Completed | 65 | 63
Not Completed | 3 | 2
Not completed — Procedure Canceled | 1 | 1
Not completed — Missed follow up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ClariFix | Sham | Total
Number analyzed (Participants) | 68 | 65 | 133
Age, Continuous [Median (Standard Deviation); unit: years] | 52.3 (15.8) | 58.3 (16.4) | 55.2 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 32 | 77
  Male | 23 | 33 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 61 | 57 | 118
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 68 | 65 | 133
Type of rhinitis (nonallergic rhinitis) [Count of Participants; unit: Participants] | 39 | 37 | 76

OUTCOME MEASURES:

1. Primary Outcome: rTNSS Responder Rate
Description: Responders are defined as participants with a 30% or greater reduction in reflective Total Nasal Symptom Score (rTNSS) relative to baseline. The active treatment will be compared with the sham treatment.
  The reflective Total Nasal Symptom Score (rTNSS) is a validated PRO consisting of 4 nasal symptom scores for rhinorrhea, nasal congestion, nasal itching, and sneezing that are assessed over the previous 2-week period. Each symptom is rated on a scale of 0 (no symptoms) to 3 (severe symptoms) and the scores are summed to provide a total rTNSS with a possible range of 0 to 12.
Time Frame: 90-days post treatment
Population: 1active ClariFix arm participant returned for the follow up visit, but did not complete the rTNSS
Measure: Count of Participants; unit: Participants
Arm/Group | ClariFix | Sham
Number analyzed (Participants) | 64 | 63
Participants | 47 | 23

2. Secondary Outcome: rTNSS Responder Rate
Description: Mean change from baseline in the rTNSS. The reflective Total Nasal Symptom Score (rTNSS) is a validated PRO consisting of 4 nasal symptom scores for rhinorrhea, nasal congestion, nasal itching, and sneezing that are assessed over the previous 2-week period. Each symptom is rated on a scale of 0 (no symptoms) to 3 (severe symptoms) and the scores are summed to provide a total rTNSS with a possible range of 0 to 12.
Time Frame: Through 12 months post treatment
Reporting Status: Not Posted, anticipated posting 2025-12

3. Secondary Outcome: Change in Total RQLQ(S)
Description: Mean change from baseline in the Standardized Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ(S)) score.
  The RQLQ(S) is a validated PRO that measures functional impairments due to allergic or non-allergic rhinoconjunctivitis. The assessment consists of 28 questions related to nose symptoms, eye symptoms, non-eye/nose symptoms, sleep problems, practical problems, activity limitations, and emotional function. Each item is scored from 0 (no impairment) to 6 (severely impaired). An overall score is calculated from the mean of the 28 item responses. Domain scores are the mean of the item scores within that domain.
Time Frame: Through 12 months post treatment
Reporting Status: Not Posted, anticipated posting 2025-12

4. Secondary Outcome: Patient Satisfaction Questionnaire
Description: Percent of participants indicating satisfaction with the procedure outcome. The satisfaction questionnaire consists of 3 questions that the participant answers at each follow-up visit. The questions indicate whether the participant is satisfied with the procedure outcome, whether the participant would undergo the procedure again for similar results, and whether the participant would recommend the procedure to family or friends with a similar condition. For each item the participant indicates agreement/disagreement with each statement.
Time Frame: Through 12 months post treatment
Reporting Status: Not Posted, anticipated posting 2025-12

5. Secondary Outcome: Serious Device- and/or Procedure-related Adverse Events
Description: The number of participants with one or more serious adverse events that are possibly, probably, or definitely related to the ClariFix device and/or procedure.
Time Frame: Through 12 months post procedure
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: Screening through 90 days
Arm/Group | ClariFix | Sham
All-Cause Mortality (participants affected / at risk) | 33/68 | 4/65
Serious Adverse Events (participants affected / at risk) | 1/68 | 1/65
Other Adverse Events (participants affected / at risk) | 33/68 | 4/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ClariFix (N=68) | Sham (N=65)
Panic Attack (Psychiatric disorders) | 1 (1) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ClariFix (N=68) | Sham (N=65)
Pain/discomfort at treatment site (Surgical and medical procedures) | 25 (25) | 1 (1)
Other (General disorders) | 8 (8) | 3 (3)

LIMITATIONS AND CAVEATS:
Study follow up is ongoing. Only 90 day endpoints are available currently.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-20): https://cdn.clinicaltrials.gov/large-docs/05/NCT04154605/Prot_SAP_000.pdf